CLINICAL TRIAL: NCT04617249
Title: Assessment of Different Routes Median and Paramedian Anesthesia in Cesarean Section
Brief Title: Median and Paramedian Anesthesia in Cesarean Section
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Aljazeera Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: anesthesia routes
Record Dates: First submitted 2020-10-31; First posted 2020-11-05 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-10

CONDITIONS: Anesthesia

STUDY DESIGN:
Intervention Model Description: anesthesia with median route versus paramedian route
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Giving median anesthesia (Active Comparator)
  Interventions: Procedure: median anesthesia
- Giving paramedian anesthesia (Active Comparator)
  Interventions: Procedure: paramedian anesthesia

INTERVENTIONS:
Procedure: median anesthesia — giving median anesthesia
  Arms: Giving median anesthesia
Procedure: paramedian anesthesia — giving paramedian anesthesia
  Arms: Giving paramedian anesthesia

SUMMARY:
The number of cesarean sections worldwide has markedly been increasing since 1985.Intrathecal anesthesia is preferred by most anesthesiologists over general anesthesia

DETAILED DESCRIPTION:
Complications with spinal anesthesia are not common which makes it difficult to detect its incidence and one of the most serious complications is nerve injury.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-42 years
* Scheduled for elective cesarean section
* ASA II

Exclusion Criteria:

* -Age <18 years or >42 years
* ASA >II
* Emergency cesarean section

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — pregnant women undergoing CS
Enrollment: 80 (Estimated)
Dates: Start 2020-11-05 (Estimated); Primary Completion 2021-04-25 (Estimated); Study Completion 2021-05-15 (Estimated)

PRIMARY OUTCOMES:
the number of women who will have less pain | 3 days
  the number of women who will have less pain post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Mahmoud Alalfy, Study Chair — Algezeera hospitaland National Research Centre ,Egypt
Locations (1):
- Aljazeera( Al Gazeera) hospital, Giza, Egypt